CLINICAL TRIAL: NCT00001115
Title: A Pilot Study to Determine the Effect of Acyclovir Treatment for Herpes Simplex Virus (HSV) Infection on Peripheral Blood HIV Viral Load.
Brief Title: The Effect of Acyclovir Treatment of the Herpes Simplex Virus (HSV) Infection on HIV Levels in the Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: DATRI 020
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 1998-06

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: Herpes Simplex; Acyclovir; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Acyclovir

INTERVENTIONS:
Drug: Acyclovir

SUMMARY:
Part A: To evaluate the impact of HSV suppression with acyclovir ( ACV ) on HIV burden in patients with asymptomatic HSV infection and at high risk for HSV reactivation.

Part B: To characterize the change in plasma HIV RNA levels and other measures of HIV burden during and after a 10 day course of ACV treatment for acute HSV infection.

Approximately 70% of patients infected with HIV are concurrently infected with HSV. There is new evidence to suggest that HSV may act as a co-factor in HIV disease progression. This study will attempt to determine if the upregulation of HIV RNA that occurs during symptomatic HSV reactivation also occurs during asymptomatic HSV reactivation and if suppression of HSV will result in decreased levels of HIV RNA. There is a need to determine the patterns of association between HSV and HIV.

DETAILED DESCRIPTION:
Approximately 70% of patients infected with HIV are concurrently infected with HSV. There is new evidence to suggest that HSV may act as a co-factor in HIV disease progression. This study will attempt to determine if the upregulation of HIV RNA that occurs during symptomatic HSV reactivation also occurs during asymptomatic HSV reactivation and if suppression of HSV will result in decreased levels of HIV RNA. There is a need to determine the patterns of association between HSV and HIV.

Part A: 60 approved HIV infected patients will be randomized to either suppressive ACV therapy or matching placebo for 12 weeks. Serology for HSV serum antibodies will be obtained at screening and a full history and physical exam will be performed on Day 1 and interval examinations at Weeks 2, 4, 8 and 12. Extensive clinical exams will be conducted on a regular schedule throughout the 12 weeks.

Part B: 15 approved HIV infected patients will receive treatment with ACV until resolution of the lesion. All patients will be monitored on Day 9-12 of ACV therapy for crusting and resolutions of HSV lesions and will be followed for 3.5 months.

AS PER AMENDMENT 3/11/97: Noncommercial active acyclovir will be made available for Part A patients wo develop acute HSV while on study and for Part B patients who develop acute HSV after completion of the acute phase of treatment ( i.e., during the follow-up phase).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

Parts A and B:

* Documented HIV infection.
* Patients >= 18 years of age must be willing and able to give informed consent and patients < 18 years must have written consent from a parent or guardian.

Part A:

* CD4+ T count < 250 cells/mm3 within 1 month prior to study entry.
* Documented antibodies to HSV any time prior to study.
* History of HSV outbreak in past 2 to 12 months.
* Former Part B patients who have completed the 12 week follow up may enter Part A after at least a 4-week washout.

Part B:

* Documented CD4+ T count < 250 cells/mm3 anytime prior to study entry.
* Oral, genital or anorectal lesions with a vesiculopustular component.
* Presumptive diagnosis of HSV.
* Former part A patients may enter part B after a 4-week washout.

Exclusion Criteria

Patients with any of the following prior conditions are excluded:

* Documented or suspected HSV within 2 months prior to study entry.
* History of infection with an acyclovir resistant HSV strain.
* History of disseminated HSV.
* History of treatment for acute CMV or MAC disease.
* History of poor medication or clinic visit compliance.

Prior Medication:

Excluded:

* Use of acyclovir, famciclovir, foscarnet, ganciclovir, valacyclovir or cidofovir for any reason within one month prior to study entry. [AS PER AMENDMENT 1/21/97: Use of antiherpes agents, both FDA-approved and investigational, including bis-POM, PMEA, lobucavir, acyclovir, etc.]
* Initiation or modification of antiretroviral therapy, immunomodulators, or any kind of vaccination within 2 months prior to study entry.
* Treatment for acute medical condition within 4 weeks prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cohn J, Study Chair; Mole L, Study Chair
Locations (15):
- United States (15):
  - AIDS Research Ctr, Palo Alto, California
  - Harbor-UCLA Med Ctr, Torrance, California
  - Yale Univ School of Medicine / AIDS Program, New Haven, Connecticut
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Illinois - Chicago, Chicago, Illinois
  - Univ of Illinois Chicago / Howard Brown Hlth Ctr, Chicago, Illinois
  - Johns Hopkins Univ, Baltimore, Maryland
  - SUNY Brooklyn / SUNY Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Community Research Initiative on AIDS, New York, New York
  - NYU - Bellevue Hosp, New York, New York
  - New York Med College / Westchester County Med Ctr, Valhalla, New York
  - Research and Education Group, Portland, Oregon
  - Univ of Pennsylvania Med Ctr, Philadelphia, Pennsylvania
  - Brown Univ / The Miriam Hosp, Providence, Rhode Island